CLINICAL TRIAL: NCT04246541
Title: Ketorolac as an Adjuvant Agent for Postoperative Pain Control Following Arthroscopic Meniscus Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Michael Karns, MD., Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20181100
Record Dates: First submitted 2020-01-24; First posted 2020-01-29 (Actual); Results first posted 2021-12-01 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Meniscus Tear, Tibial; Pain, Postoperative; Postoperative Complications; Ketorolac Adverse Reaction; Opioid Use
Keywords: ketorolac; meniscus tear; analgesics; pain
MeSH Terms: conditions — Tibial Meniscus Injuries; Pain, Postoperative; Postoperative Complications; Pain | interventions — Ketorolac; oxycodone-acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Experimental): Patients will receive standard of care Percocet for post-operative pain control following meniscus debridement surgery
  Interventions: Drug: Oxycodone-Acetaminophen
- Ketorolac (Experimental): Patients will receive IV ketorolac during surgery. They will then receive 3 days of oral ketorolac every 6 hours for pain control following surgery.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — Patients will receive IV ketorolac during surgery followed by 3 days of oral ketorolac (10 mg every 6 hours) for pain control. Patients will also be given oxycodone-acetaminophen (5mg-325mg) PRN for pain not controlled with ketorolac.
  Arms: Ketorolac
Drug: Oxycodone-Acetaminophen — Patients will be discharged with oxycodone-acetaminophen (5mg-325mg) PRN for pain control after surgery.
  Arms: Control

SUMMARY:
The utilization of arthroscopic surgery to treat meniscus injuries has continued to increase in recent years, partly due to a younger, more active population, and improved technology and technique. However, pain management in the post-operative period is critical to the ability to perform this procedure as an outpatient surgery. Traditionally, oral narcotic agents have been the preferred analgesic postoperatively in orthopaedic surgery. However, these agents are associated with several side effects, including nausea/vomiting, constipation, and somnolence. In addition, opioid agents have a significant potential for abuse in comparison to non-narcotic analgesics. In light of the rising opioid epidemic and nationwide initiatives to limit narcotic usage, surgeons must explore alternate pain modalities in the acute postoperative period. Ketorolac is a non-steroidal anti-inflammatory drug (NSAID) with analgesic and anti-inflammatory properties.1 Multiple prior studies have examined the beneficial effect of oral and intravenous (IV) ketorolac as an analgesic in the postoperative period,1-3 including arthroscopic meniscus surgery. However, the beneficial effects of this agent following arthroscopic meniscus surgery have not been extensively described.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 89 years of age
* Patients undergoing primary arthroscopic meniscus surgery

Exclusion Criteria:

* Patients age less than 18 or greater than 89 years
* Illiterate or non-English speaking patients
* Patients with contraindications to ketorolac
* History of drug or alcohol abuse
* Chronic use of analgesic or psychotropic drugs

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Karns, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- UH Cleveland Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Ketorolac
Started | 25 | 23
Completed | 22 | 20
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Ketorolac | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 23 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (15.6) | 47.9 (13.1) | 47.9 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 12 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 25 | 23 | 48
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Pain Levels Recorded With a Visual Analogue Scale
Description: Patients will record pain levels post-operatively using a visual analogue scale (VAS) ranging from 0 as the minimum value to 100 as the maximum value. A smaller VAS value will be considered a lower pain level.
Time Frame: 2 weeks postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 25 | 23
score on a scale | 25.6 (22.7) | 28.8 (26.3)

2. Primary Outcome: Narcotic Medication Consumed
Description: Number of oxycodone- acetaminophen tablets consumed
Time Frame: up to 5 days postoperatively
Population: 9 subjects, including 4 in the control group and 5 in the ketorolac group, failed to report complete data on postoperative number of oxycodone-acetaminophen tablets consumed and were therefore excluded from data analysis.
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 21 | 18
tablets | 5.7 (7.2) | 3.5 (3.7)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Control | Ketorolac
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23

LIMITATIONS AND CAVEATS:
single institution study not blinded

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT04246541/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/41/NCT04246541/ICF_001.pdf